CLINICAL TRIAL: NCT04191668
Title: A Validation Study of the NightOwl PAT-based Home Sleep Apnea Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ectosense NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NightOwl-01
Record Dates: First submitted 2019-11-19; First posted 2019-12-10 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Single Group will undergo both gold standard polysomnography (PSG) and NightOwl Sleep Apnea Test
Masking Description: Sleep technician which analyses the PSG data will be blinded from any prior PSG analysis and the NightOwl analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PSG and NightOwl (Other): Default patient recruitment During the study, for each execution day, all patients that have been scheduled for a PSG will be presented with an informed consent. All recruited patients shall be a part of the study during which they wear the NightOwl Sensor while undergoing the PSG exam.
  Interventions: Device: NightOwl

INTERVENTIONS:
Device: NightOwl — The NightOwl is a finger-mounted home sleep apnea testing device

SUMMARY:
The objective of this study is to evaluate the performance of a miniaturized sleep apnea test, called NightOwl. The system consists of a sensor placed on the fingertip and a cloud-based analytics software. The sensor acquires accelerometer and photoplethysmographic data. The software derives actigraphy from the former, and blood oxygen saturation and peripheral arterial tone (PAT), among other features, from the latter. In order to assess NightOwl's performance, the investigators will compare the respiratory event index (REI), defined as the number of respiratory events per hour of sleep, derived by the NightOwl system, to the apnea-hypopnea index (AHI) obtained from manual analysis of the polysomnography (PSG), which is the gold standard for sleep apnea diagnosis. The investigators will also compare the total sleep time (TST) derived by both systems. This study will be performed in a sleep lab environment.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the performance of a miniaturized sleep apnea test, called NightOwl. The system consists of a sensor placed on the fingertip and a cloud-based analytics software. The sensor acquires accelerometer and photoplethysmographic data. The software derives actigraphy from the former, and blood oxygen saturation and peripheral arterial tone (PAT), among other features, from the latter. In order to assess NightOwl's performance, The investigators will compare the respiratory event index (REI), defined as the number of respiratory events per hour of sleep, derived by the NightOwl system, to the AHI obtained from manual analysis of the polysomnography (PSG), which is the gold standard for sleep apnea diagnosis. The investigators will also compare the total sleep time (TST) derived by both systems. This study will be performed in a sleep lab environment.

As of March 2017, the new clinical practice guideline for diagnostic testing for adult sleep apnea of the American Academy of Sleep Medicine (AASM) for the first time formulates a strong recommendation that both polysomnography (PSG) and home sleep apnea testing (HSAT) are appropriate diagnostic testing options for uncomplicated adult patients who are at increased risk of moderate to severe sleep apnea.

Collop et al. performed a comprehensive analysis of the evidence for HSAT devices to diagnose obstructive sleep apnea (OSA) in out-of-center settings. The authors concluded that testing devices that analyze changes in peripheral arterial tone (PAT) in combination with actigraphy and blood oxygen saturation (SpO2) are adequate to diagnose OSA in patient populations with a high pre-test probability.

In this study, the investigators wish to assess the performance of a system for the diagnosis of OSA that measures and analyzes the abovementioned parameters, called NightOwl. The system consists of a small sensor device which is placed on the fingertip and a cloud-based analytics platform.

It is designed to be self-applied and initiated by the patient by attaching the sensor to the fingertip by means of an adhesive patch.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an indication for an in-lab polysomnography

Exclusion Criteria:

* Intellectually disabled people
* People younger than 13 years of age.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Massie, MSc, Study Director — Ectosense NV
Locations (3):
- United States (3):
  - Miami Lakes Laboratory, Miami Lakes, Florida
  - Plantation Laboratory East, Plantation, Florida
  - Plantation Laboratory West, Plantation, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Massie F, Vits S, Verbraecken J, Bergmann J. Context-aware analysis enhances autoscoring accuracy of home sleep apnea testing. J Clin Sleep Med. 2025 May 1;21(5):789-804. doi: 10.5664/jcsm.11534. PMID 39748512
- [Derived] Van Pee B, Massie F, Vits S, Dreesen P, Klerkx S, Bijwadia J, Verbraecken J, Bergmann J. A multicentric validation study of a novel home sleep apnea test based on peripheral arterial tonometry. Sleep. 2022 May 12;45(5):zsac028. doi: 10.1093/sleep/zsac028. Epub 2022 Feb 2. PMID 35554589

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PSG and NightOwl
Started | 106
Completed | 106
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only participants for which technically adequate polysomnography and home sleep apnea test data was acquired were retained for Baseline Analysis
Arm/Group | PSG and NightOwl
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For one participant, gender data could not be retrieved.
  Participants
    number analyzed (Participants) | 72
    Female | 42
    Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 18
  Race: White | 54
  Race: Not reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 73
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.6 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Pearson Correlation Between the AHI
Description: The evaluation of the Pearson correlation between the apnea-hypopnea index (AHI) estimate obtained from the NightOwl and the AHI determined from the polysomnography (PSG); The AHI is defined as the number of apnea or hypopnea divided by the (estimated) total sleep time expressed in hours.
Time Frame: Through study completion, an average of 1 month.
Population: The population comprised those participants for which technically adequate polysomnography and home sleep apnea test data could be acquired.
Measure: Number; unit: Correlation coefficient
Arm/Group | PSG and NightOwl
Number analyzed (Participants) | 73
Correlation coefficient | 0.909

2. Primary Outcome: Pearson Correlation Between the TST
Description: The evaluation of the Pearson correlation between the total sleep time (TST) estimate obtained from the NightOwl and the TST determined from the PSG;
Time Frame: Through study completion, an average of 1 month.
Population: as for outcome 1
Measure: Number; unit: Correlation coefficient
Arm/Group | PSG and NightOwl
Number analyzed (Participants) | 73
Correlation coefficient | 0.610

3. Primary Outcome: The Evaluation of the Level of Agreement (Classification Accuracy) Between Patient Categorization
Description: The evaluation of the level agreement (classification accuracy) between patient categorization (into sleep apnea severity categories) obtained by the NightOwl and those obtained by the PSG. This measure is calculated by dividing the number of participants on which both NightOwl and the PSG agree on the sleep apnea severity category by the total number of participants.
Time Frame: Through study completion, an average of 1 month.
Population: as for outcome 1
Measure: Number; unit: Ratio
Arm/Group | PSG and NightOwl
Number analyzed (Participants) | 73
Ratio | 0.685

ADVERSE EVENTS:
Time Frame: Through study completion (during the participant's single-night sleep study)
Arm/Group | PSG and NightOwl
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT04191668/Prot_SAP_000.pdf